CLINICAL TRIAL: NCT00223262
Title: Clinical Trial of Lamotrigine to Reverse Cognitive Impairment in Chronic Corticosteroid-Treated Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sherwood Brown, UT Southwestern Medical Center at Dallas
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: LMC-R62
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Memory Impairment Due to Corticosteroid Use; Hypomania Due to Corticosteroid Use; Hippocampal Atrophy Due to Corticosteroid
MeSH Terms: interventions — Lamotrigine; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Lamotrigine (Drug)

SUMMARY:
The purpose of this study is to determine if lamotrigine therapy is associated with improvement in mood, memory and hippocampal size and function in patients receiving chronic corticosteroid therapy. Standard care for mood changes associated with corticosteroid therapy, if severe, includes antidepressants or other medications which can influence mood. No therapies, other than dose reduction or discontinuation, are currently available for memory loss associated with corticosteroid treatment. However, very little information is available on the treatment of either mood or memory changes associated with corticosteroid treatment, thus the proposed project may improve standard care.

ELIGIBILITY:
Inclusion Criteria:

* Current Corticosteroid Use of 7 mg or more for 6+ months
* 18-65 years of age

Exclusion Criteria:

* Primarily non-English speaking
* Pregnant/nursing woman
* Currently taking Depakote
* Currently taking Rifampin
* Has diagnosis of major depressive disorder, schizophrenia, PTSD, bipolar I or bipolar II (not related to corticosteroid use)
* Diseases with CNS involvement
* Is to start a brief steroid taper
* History of Alcohol/drug abuse/dependence

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2002-08; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, Ph.D., M.D., Principal Investigator — The UT Southwestern Medical Center
Locations (1):
- The UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lamotrigine: Lamotrigine was initiated at 25 mg/day for 2 weeks, increased to 50 mg/day for 2 weeks, and then increased in 50 mg/day increments weekly to a dose of 400 mg/day at week 10 using a fixed dosing schedule.
- Placebo: Matched placebo identical in appearance to the active drug.
Period: Overall Study
Arm/Group | Lamotrigine | Placebo
Started | 16 | 12
Completed | 8 | 11
Not Completed | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamotrigine | Placebo | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (11.2) | 47.4 (13.3) | 46.0 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Rey Auditory Verbal Learning Test (RAVLT)
Description: Rey Auditory Verbal Learning Test (RAVLT) is a test of verbal learning and declarative memory. During the test, 15 nouns that are read aloud for 5 consecutive trials. Each trial is followed by a free recall test (participant is asked to recall the words that were just read to them). The sum of correctly recalled words across 5 trials is called the total raw score. On completion of Trial 5, an interference list of 15 words (List B) is presented, followed by a free recall test of that list. After a 20-min delay, the examinee is again required to recall the words from list A - this is called the delay raw score. The raw scores on both the total recall and the delay trials (number of words correct across trials 1-5) are converted to standardized T-scores (Mean=50; SD=10; range 20-100) based on participant age and gender. The scores below are presented as T-scores, with higher scores indicative of better performance.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 8 | 11
T-scores | 46.1 (15.0) | 40.1 (11.0)

ADVERSE EVENTS:
Arm/Group | Lamotrigine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/8 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No